CLINICAL TRIAL: NCT06292312
Title: Investigation of the Effectiveness of Craniosacral Therapy in Patients With Multiple Sclerosis: A Randomized Controlled, Single-Blind Study
Brief Title: Investigation of the Effectiveness of Craniosacral Therapy in Patients With Multiple Sclerosis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Lokman Hekim University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19.12.2023/10-483
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; craniosacral therapy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: dual parallel group design
Who Masked: Outcomes Assessor
Masking Description: Single (outcomes assesor) The evaluation of the patients will be carried out by a blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Patients in this grop are the group to which craniosacral therapy and convensional physiotherapy will be applied.
  Interventions: Other: Craniosacral therapy; Other: Conventional physiotherapy
- Control group (Active Comparator): Patients in this group are the group to which conventional physiotherapy will be applied.
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Other: Craniosacral therapy — Craniosacral therapy is defined as an alternative, massage-like treatment approach using gentle manual force to address somatic dysfunctions of the head and the rest of the body.
  Other Names: Conventional physiotherapy
  Arms: Treatment group
Other: Conventional physiotherapy — Range of motion, stretching, resistance exercises. Spasticity inhibition Balance and coordination exercises Walking training Stabilization exercises Breathing exercises

SUMMARY:
Although the cause of Multiple Sclerosis (MS), one of the common demyelinating diseases of the central nervous system, has not yet been fully elucidated, autonomic nervous system dysfunction has been suggested in its etiology. Symptoms such as fatigue, problems with bladder, bowel, cardiovascular, sleep, sexual and sweating functions, abnormal sympathetic skin response or decreased heart rate variation support this hypothesis.

In the treatment of many neurological diseases such as Multiple Sclerosis, complementary medicine practices and non-traditional therapies have recently been shown to be effective in addition to conventional practices. One of these practices, craniosacral therapy (CST), uses manual palpation and manipulation of the craniosacral system to influence sensory, motor, cognitive and emotional processes in the nervous system. In addition, it is thought that applying external force to certain bone elements can have a positive effect on various symptoms in patients with MS, based on the knowledge that it can be transmitted within the system.

DETAILED DESCRIPTION:
In addition to pharmacological treatments, many non-pharmacological treatment modalities such as physiotherapy applications, sleep hygiene training, relaxation techniques, behavioral therapy and cognitive therapies are used in the treatment of MS symptoms. Recently, complementary medicine practices and non-traditional therapies have been shown to be effective in the treatment of many neurological diseases, including MS. Among these methods, craniosacral therapy (CST) has been shown to be effective in the treatment of various neurological conditions affecting the central nervous system. CST is defined as an alternative, massage-like treatment approach using gentle manual force to address somatic dysfunctions of the head and the rest of the body. The interplay of diagnosis and treatment aims to mobilize cranial sutures that abnormally restrict physiological movement.

CST is an approach widely used in adults and children, in different clinical settings and conditions. Based on the knowledge that the application of external force to certain bony elements of this system can be transmitted within the system, it can be considered that craniosacral therapy may have a positive effect on various symptoms in patients with MS. In the light of the results obtained as a result of the study, CST may provide ideas to clinicians and researchers as an alternative and complementary method in the treatment of MS.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* Definitive diagnosis of MS by a neurologist
* EDSS score between 1-5.5
* Not receiving active physical therapy services
* Volunteering.

Exclusion Criteria:

* Having a neurological disease other than MS
* Attacks in the last three months
* Corticosteraoid use
* History of surgery on the spine
* Central and peripheral nervous system disease
* Pregnancy
* Oncological diseases
* Severe comorbid somatic and psychiatric disorders
* Receiving invasive/manipulative treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Dynamic posturography | Change from baseline at 8 weeks treatment program and two months after.
  Dynamic posturography is a device that converts the balance of the individual under changing floor, environment and stimulus conditions into computerized data with receivers on the floor.
Heart rate variability | Change from baseline at 8 weeks treatment program and two months after.
  Heart rate variability is a tool that allows the investigation of cardiovascular autonomic function through the measurement of variations in RR intervals and provides valuable information about the control of autonomic nervous system.
Number of participants | Change from baseline at 8 weeks treatment program and two months after.
  A total of 32 MS patients, 16 in both groups, will be included in the study.

SECONDARY OUTCOMES:
Pain level | Change from baseline at 8 weeks treatment program and two months after.
  Visual analog scale will be used to examine pain levels of participants. Individuals are presented with a line numbered evenly from 1 to 10 and asked to mark the point corresponding to their pain intensity. A higher score indicates that severity of pain increasing.
Central sensitization | Change from baseline at 8 weeks treatment program and two months after.
  The Central Sensitization Scale (CSS) will be used. The CSS was developed as a screening tool to better assess symptoms thought to be associated with CS, categorize syndromes, define disease severity, measure sensitivity, and assist physicians and clinicians in treatment planning by minimizing or, if possible, avoiding unnecessary diagnostic and treatment procedures. Part A of the SSI includes all CS symptoms and is the part that will help clinicians to recognize the CS patient. According to the scale, those with a score above 40 are considered to have developed CS.
Fatigue | Change from baseline at 8 weeks treatment program and two months after.
  Fatigue Severity Scale will be applied. Each item in the self-administered 9-question scale, which reflects the situation of the individuals in the last week, consists of "1" Strongly disagree, "7" It consists of a score between "1-7" corresponding to the statement "I agree". As a result of dividing the total score obtained by the number of questions, ">6.1" corresponds to chronic fatigue syndrome and "<2.8" to no fatigue. The lower the total score, the less fatigue is interpreted
Sleep quality | Change from baseline at 8 weeks treatment program and two months after.
  Pittsburgh Sleep Quality Index (PSQI) will be used. The PSQI is a self-report scale that assesses sleep quality and sleep disturbance over a one-month period. The PDQI has 7 components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, sleep medication use and daytime dysfunction. Some of the components are indicated by a single item, while others are obtained by grouping several items. Each item is evaluated on a 0-3 point scale and the sum of the 7 component scores constitutes the total PDQI score. The total score has a value between 0-21, with a high total score indicating poor sleep quality.
Life quality | Change from baseline at 8 weeks treatment program and two months after.
  Multiple Sclerosis Quality of Life Scale (MSQoL-54) scale will be used. It was created by Vickrey et al. (1995) by adding 18 items specific to MS to the SF-36 quality of life scale used in many diseases. The MSQoL was created by adding 18 items to the items in the SF-36 related to general health perception (5 items), energy/fatigue (4 items), social function (2 items), emotional flexibility (5 items), limitations due to emotional problems (3 items), limitations due to physical problems (4 items), physical function (10 items), pain (2 items) and change in health. The 2 main groups of the scale score between 0-100, with higher scores indicating higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Aslan, MSc, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Indivudual participant data will be available to the responsible researcher.